CLINICAL TRIAL: NCT04012268
Title: The Safety and Effect of Remote Ischemic Conditioning on Adult Moyamoya Disease
Brief Title: The Safety and Efficacy of RIC on Adult Moyamoya Disease
Acronym: RIC-AMD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Ji Xunming,MD,PhD, Professor, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RIC-AMD
Record Dates: First submitted 2019-07-03; First posted 2019-07-09 (Actual); Last update posted 2021-03-12 (Actual); Status verified 2021-03

CONDITIONS: Moyamoya Disease
Keywords: moyamoya disease; remote ischemic conditioning; cerebral blood flow
MeSH Terms: conditions — Moyamoya Disease | interventions — Aspirin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RIC group (Experimental): Patients allocated to the RIC group will undergo RIC procedure during which bilateral arm cuffs are inflated to a pressure of 50 mmHg over systolic blood pressure for five cycles of 5 min followed by 5 min of relaxation of the cuffs. They will also accept medication treatment by professional neurologists.
  Interventions: Device: RIC
- Medication group (Other): Patients allocated to Medication group will accept medication treatment by professional neurologists.
  Interventions: Drug: Aspirin

INTERVENTIONS:
Device: RIC — Patients allocated to the RIC group will undergo RIC procedure during which bilateral arm cuffs are inflated to a pressure of 50 mmHg over systolic blood pressure for five cycles of 5 min followed by 5 min of relaxation of the cuffs.
  Arms: RIC group
Drug: Aspirin — patients will accept medication guided by neurologists
  Arms: Medication group

SUMMARY:
There are a series of symptoms such as ischemic stroke、transient ischemic attack 、hemorrhagic stroke、headache 、seizure and so on in moyamoya disease( MMD) patients .Nowadays, revascularization is the only effective way for ischemic MMD and there is no effective conservative treatment for MMD. This study was to explore the safety and efficacy of remote ischemic conditioning(RIC ) on adult MMD patients.

DETAILED DESCRIPTION:
There are a series of symptoms such as ischemic stroke、transient ischemic attack 、hemorrhagic stroke、headache 、seizure and so on in moyamoya disease. Nowadays, revascularization is the only effective way for ischemic MMD while controversial for hemorrhagic MMD patients. Surgical complications including hyperperfusion syndrome, cerebral infarction or bleeding often occurred postoperatively. There is no effective conservative treatment for MMD up to now.

Remote ischemic conditioning is Remote ischemic conditioning (RIC) is a noninvasive and easy-to-use neuroprotective strategy, and it has potential effects on preventing ischemia reperfusion injury and ischemic infarction.This study was to explore the safety and efficacy of remote ischemic conditioning on adult MMD patients.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-60 years
* All of the patients underwent digital subtraction angiography (DSA) and met the current diagnostic criteria recommended by the Research Committee on MMD of the Ministry of Health and Welfare of Japan in 2012.
* mRs≤3
* Informed consent obtained from patient or acceptable patient's surrogate.

Exclusion Criteria:

* Patients with acute ischemic or hemorrhagic stroke within 3 months.
* Severe hepatic or renal dysfunction.
* Severe hemostatic disorder or severe coagulation dysfunction.
* Severe cardiac diseases.
* Patients with severe existing neurological or psychiatric disease
* Patients with moyamoya syndrome caused by autoimmune disease, Down syndrome , neurofibromatosis, leptospiral infection, or previous skull-base radiation therapy.
* Patients have been done or plan to accept revascularization surgery.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2020-11-10 (Actual); Study Completion 2021-02-02 (Actual)

PRIMARY OUTCOMES:
improvement ratio of mean cerebral blood flow | change from the baseline to12 months after treatment
  Cerebral blood flow refers to the flow of blood through a certain cross-sectional area of cerebrovascular in a unit time. Patients' CBF will be detected by arterial spin labeling. In each hemisphere, middle cerebral artery territory was divided into ten regions according to Albert Stroke Program Early CT score (ASPECTS), regions of interest (ROI) were drawn manually in each of territory of MCA to determine the absolute CBF values. improvement ratio of mean CBF= mCBF atter treatment-mCBF baseline/mCBF baseline.

SECONDARY OUTCOMES:
incidence of ischemic stroke | from the baseline to 12 months after treatment
  ischemic stroke is diagnosed by symptoms of neurologic deficit or head CT and MRI.
incidence of transient ischemic attack | from the baseline to 12 months after treatment
  TIA is diagnosed by patients' transient neurologic deficit
incidence of hemorrhagic stroke | from the baseline to 12 months after treatment
  hemorrhagic stroke is diagnosed by head CT
The level of matrix metalloproteinase 9 (MMP-9) | change from the baseline to 3, 6, 12 months after treatment
  Blood samples will be drawn from cubital vein to test these biomarkersThese samples will be centrifuged immediately after collection and stored at - 80 until batch evaluation
The level of vascular endothelial growth factor | change from the baseline to 3, 6, 12 months after treatment
  Blood samples will be drawn from cubital vein to test these biomarkersThese samples will be centrifuged immediately after collection and stored at - 80 until batch evaluation
The level of basic fibroblast growth factor | change from the baseline to 3, 6 ,12 months after treatment
  Blood samples will be drawn from cubital vein to test these biomarkersThese samples will be centrifuged immediately after collection and stored at - 80 until batch evaluation
The rate of death and adverse event | change from the baseline to 12 months after treatment
  All causes of death will be included to compute mortality at 12 months after therapy
The number of patients with erythema,and/or skin lesions related to RIC | change from the baseline to 12 months after treatment
  Professional doctors will check it and the investigator will record the number.
The number of patients not tolerating RIC procedure,and refuse to continue the RIC procedure | change from the baseline to 12 months after treatment
  the investigator will record the number.
The rate of progression of stenosis or occlusion at Willis circle | 12 months after therapy
  Progression of stenosis or occlusion at Willis circle was evaluated by TOF-MRA, which was defined as the the stenosis or occlusion was progressed to another part of Willis circle, like stenosis progressed from M1 to M2-M4 et al, or in the same part, stenosis progressed to occlusion.

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, Beijing Municipality, China